CLINICAL TRIAL: NCT02645838
Title: Motivational Interviewing Versus Brief Advice for Smoking Cessation in General Practice
Brief Title: Motivational Interviewing for Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Yafang Huang, MD, PHD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CMUGP
Record Dates: First submitted 2015-12-24; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Smoking Cessation
Keywords: Motivational Interviewing; Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing group (Experimental): 1. Structural motivational interviewing for one section (about 20 mins)，provided by family physician
  2. Follow-up telephone call，provided by family physician
  Interventions: Behavioral: Motivational interviewing
- Brief advice group (No Intervention): Brief advice without motivational interviewing (about 5 mins), provided by family physician

INTERVENTIONS:
Behavioral: Motivational interviewing — 1. Structural motivational interviewing for one section (about 20 mins)，provided by family physician;2. Follow-up telephone call，provided by family physician.
  Arms: Motivational interviewing group

SUMMARY:
The purpose of this study is to determine whether or not motivational interviewing is effective in smoking cessation at general practice setting in China.

DETAILED DESCRIPTION:
OBJECTIVES:

• To compare the effectiveness of motivational interviewing versus brief advice by conducting a randomized controlled trial in General Practice Setting in China.

OUTLINE:

This is a randomized controlled study. Patients are randomized to either the intervention arm or the control arm.

• Arm I (intervention): Patients will be given a 20 minutes personal talk in the family physician's office during the visit. The family physicians will determine the stage of change in smoking cessation (precontemplative, contemplative, action, maintenance and relapse) and use the motivational interviewing skills during the talk. The motivational interviewing skills include expressing empathy, developing discrepancy, rolling with resistance, supporting self efficacy. Up to six phone calls will be given to the patients during the follow-up, using the motivational interviewing skill.

• Arm II (control): Patients will receive brief advice for smoking cessation, lasting approximately 5 minutes. The risks of smoking and the advantages of quitting will be explained. The information provided during the talk will be standardized. No phone call will be given during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 80 years.
2. Any person who replies "Yes" when asked "Do you smoke?".
3. Agree to participate the trial and be followed for at least one year.

Exclusion Criteria:

1. With severe mental illness, serious drug dependent patients.
2. Cannot understand conversation or cannot communicate, such as deafness or dementia.
3. Cannot be followed up for one year, such as not likely survive for more than one year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
1 week point prevalence abstinence (PPA) | Self-reported PPA at 1 week follow-up
  Validation: exhaled carbon monoxide (CO) (< 10 ppm)

SECONDARY OUTCOMES:
1 month PPA | Self-reported 7-day PPA at 1 month follow-up
  Validation: exhaled CO (< 10 ppm)
3 month PPA | Self-reported 7-day PPA at 3 month follow-up
  Validation: exhaled CO (< 10 ppm)
6 month PPA | Self-reported 7-day PPA at 6 month follow-up
  Validation: exhaled CO (< 10 ppm)

CONTACTS AND LOCATIONS:
Overall Officials: Yafang Huang, PHD, Principal Investigator — School of General Practice and Continuing Education, Capital Medical University

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be available.

REFERENCES:
- [Background] Bock BC, Papandonatos GD, de Dios MA, Abrams DB, Azam MM, Fagan M, Sweeney PJ, Stein MD, Niaura R. Tobacco cessation among low-income smokers: motivational enhancement and nicotine patch treatment. Nicotine Tob Res. 2014 Apr;16(4):413-22. doi: 10.1093/ntr/ntt166. Epub 2013 Oct 30. PMID 24174612
- [Background] Borrelli B, Novak S, Hecht J, Emmons K, Papandonatos G, Abrams D. Home health care nurses as a new channel for smoking cessation treatment: outcomes from project CARES (Community-nurse Assisted Research and Education on Smoking). Prev Med. 2005 Nov-Dec;41(5-6):815-21. doi: 10.1016/j.ypmed.2005.08.004. Epub 2005 Sep 22. PMID 16182355
- [Background] Davis MF, Shapiro D, Windsor R, Whalen P, Rhode R, Miller HS, Sechrest L. Motivational interviewing versus prescriptive advice for smokers who are not ready to quit. Patient Educ Couns. 2011 Apr;83(1):129-33. doi: 10.1016/j.pec.2010.04.024. PMID 20627440
- [Background] Glasgow RE, Whitlock EP, Eakin EG, Lichtenstein E. A brief smoking cessation intervention for women in low-income planned parenthood clinics. Am J Public Health. 2000 May;90(5):786-9. doi: 10.2105/ajph.90.5.786. PMID 10800431
- [Background] Mantler T, Irwin JD, Morrow D. Motivational interviewing and smoking behaviors: a critical appraisal and literature review of selected cessation initiatives. Psychol Rep. 2012 Apr;110(2):445-60. doi: 10.2466/02.06.13.18.PR0.110.2.445-460. PMID 22662398
- [Background] Miller RW, Rollnick S. Motivational Interviewing: Preparing people to change addictive behavior. New York: Guilford Press; 1991.